CLINICAL TRIAL: NCT07224685
Title: Evaluation of Voice and ECG Transmission and AI Models Using Voice, ECG and Health Data Collected Using a Mayo Clinic Center for Digital Health (CDH)-Developed App for a Repository: Mayo Clinic CV Research for Heart & Voice Study
Brief Title: A Study of Mayo Clinic CV Research Heart & Voice Study
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Paul A. Friedman, Principal Investigator, Mayo Clinic
Other Study IDs: 23-012146
Record Dates: First submitted 2025-11-03; First posted 2025-11-05 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-10

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients using the Mayo patient iPhone app
  Interventions: Other: Voice Recording

INTERVENTIONS:
Other: Voice Recording — Patients will record a 30-second to 2-minute video pronouncing vowel sounds or reading a short script. This will occur every 14 days for up to five years.

SUMMARY:
The purpose of the study is to determine whether voice recordings acquired from patient-owned Android and Apple (iOS) smartphones can be used to monitor cardiovascular health. Voice signals will be processed to determine whether we can detect presence of cardiovascular disease and wellness, or if health risks exist.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients using the Mayo patient iPhone app and iOS 14.0 or later (determined automatically via Mayo software) and Apple Watch v 4 or later (not SE), or if they have Android device for voice
* Expressed interest in participation
* Signed HIPPA authorization

Exclusion Criteria:

• Age under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who have the Mayo Clinic app and iOS 14 or Android smartphone (other types of smartphones will be added when functionality is added to the CDH app).
Sampling Method: Non-Probability Sample
Enrollment: 1000000 (Estimated)
Dates: Start 2024-03-05 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Total Patients Who Recorded a Voice Sample | Baseline
  The total number of patients who recorded a voice sample will be defined as those completing a 30-second to 2-minute video, pronouncing vowel sounds or reading a short script as prompted by the Mayo Clinic App.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Friedman, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No